CLINICAL TRIAL: NCT04949555
Title: Long Term Evaluation of Primary Congenital Glaucoma Management In Sohag University Hospital
Acronym: PCG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ghada Fathy Mohamed, resident practitioner of ophthalmology.principal investigator, Sohag University
Other Study IDs: SohajuGF
Record Dates: First submitted 2021-06-16; First posted 2021-07-02 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Primary Congenital Glaucoma
Keywords: primary congenital glaucoma
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Primary congenital glaucoma evaluation — long term evaluation of primary congenital glaucoma management

SUMMARY:
evaluation of primary congenital glaucoma management in sohag university hospital

DETAILED DESCRIPTION:
long term evaluation of primary congenital glaucoma management in sohag university hospital

ELIGIBILITY:
Inclusion Criteria:

* children operated more than 3 months

Exclusion Criteria:

* other types of operated pediatric glaucoma

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient s with primary congenital glaucoma operated in sohag university hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of patient with primary congenital glaucoma managed in sohag university hospital by surgical intervention,trabeculectomy and trabecultomy with mitomycin and ologen.follow up after management by measuring intra ocular pressure by Perkins. | 3years
  retrospective study

CONTACTS AND LOCATIONS:
Overall Officials: ghada f mohamed, MBBCH, Principal Investigator — Sohag University
Locations (1):
- Ghada Fathy Mohamed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT04949555/Prot_000.pdf